CLINICAL TRIAL: NCT04745260
Title: A Randomized Controlled Trial of Intranasal Fentanyl in Combination With Midazolam Versus Midazolam Alone for Analgesia and Anxiolysis During Pediatric Facial Laceration Repair
Brief Title: Intranasal Fentanyl in Combination With Midazolam Versus Midazolam Alone for Pediatric Facial Laceration Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Brittany DiFabio, Pediatric Emergency Medicine Fellow Physician, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020040016
Record Dates: First submitted 2021-01-31; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Facial Laceration; Anxiety
Keywords: Laceration repair; Facial laceration; Anxiety; Midazolam; Fentanyl
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A non-blinded researcher (physician) will determine the group to which the patient is assigned and order the medication(s) according to the assigned group. A separate blinded researcher (physician) will then perform the laceration repair, mYPAS, and post-procedure evaluations. The non-blinded researcher, nurse, parent, and patient will be advised not to disclose which medication(s) were administered to ensure blinding of the provider performing the laceration repair and assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intranasal Midazolam and Intranasal Fentanyl (Experimental): Study participants assigned to the combination (experimental) group will receive a weight-based dose of intranasal Fentanyl (50mcg/mL concentration at 2mcg/kg up to 100mcg) followed by intranasal Midazolam (5mg/mL concentration at 0.2mg/kg up to 10mg) using a mucosal atomizer device (1mL syringe with an attached atomizer).
  Interventions: Drug: Intranasal Fentanyl Spray and Intranasal Midazolam Spray
- Intranasal Midazolam (Active Comparator): Study participants assigned to the control (active comparator) group will receive only intranasal Midazolam (5mg/mL concentration at 0.3mg/kg up to 10mg) using a mucosal atomizer device (1mL syringe with an attached atomizer).
  Interventions: Drug: Intranasal Midazolam Spray

INTERVENTIONS:
Drug: Intranasal Fentanyl Spray and Intranasal Midazolam Spray — Intranasal Fentanyl 2mcg/kg and Intranasal Midazolam 0.2mg/kg
  Other Names: Versed
  Arms: Intranasal Midazolam and Intranasal Fentanyl
Drug: Intranasal Midazolam Spray — Intranasal Midazolam 0.3mg/kg
  Other Names: Versed
  Arms: Intranasal Midazolam

SUMMARY:
The purpose of the study is to compare the effectiveness of a combination of intranasal fentanyl and intranasal midazolam to intranasal midazolam alone for analgesia and anxiolysis in patients presenting for facial laceration repair in the pediatric emergency department.

DETAILED DESCRIPTION:
This study will be a single blind (blinded observer) randomized control trial to evaluate the efficacy of the combination of intranasal fentanyl and intranasal midazolam compared to intranasal midazolam alone for analgesia and anxiolysis during pediatric facial laceration repair.

ELIGIBILITY:
Inclusion Criteria:

* Facial laceration requiring repair with sutures
* English or Spanish-speaking parent/guardian

Exclusion Criteria:

* Lacerations requiring IV sedation or subspecialist involvement
* Patient has other injuries requiring medical attention
* Patient has vital sign instability, per physician discretion
* Patient has autism spectrum disorder
* Patient has allergies to either medication

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Score (mYPAS) | Pre-procedure
  mYPAS score at time of positioning, to be completed by blinded researcher (provider) to assess anxiety level. Scores range from 22.5 to 100, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Provider Satisfaction with Procedural Sedation (Visual Analog Score) | Immediately after the procedure
  VAS (visual analog score) completed by blinded researcher (provider) to rate satisfaction with level of sedation and ease of procedure. The scale will range from 0 (unsatisfied) to 100 (very satisfied).
Parent Satisfaction with Anxiolysis (Visual Analog Scale) | Immediately after the procedure
  VAS (visual analog score) completed by parent to rate satisfaction with level of anxiolysis for procedure. The scale will range from 0 (unsatisfied) to 100 (very satisfied).
Rate of Treatment Failure | Immediately after the procedure
  Failure of intervention to provide appropriate anxiolysis and need for IV sedation
Duration of Procedure | Immediately after the procedure
  Duration of procedure from positioning to last suture placement, to be recorded by blinded researcher (provider)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany J DiFabio, MD, Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fein JA, Zempsky WT, Cravero JP; Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine; American Academy of Pediatrics. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2012 Nov;130(5):e1391-405. doi: 10.1542/peds.2012-2536. Epub 2012 Oct 29. PMID 23109683
- [Background] Kennedy RM, Luhmann JD. The "ouchless emergency department". Getting closer: advances in decreasing distress during painful procedures in the emergency department. Pediatr Clin North Am. 1999 Dec;46(6):1215-47, vii-viii. doi: 10.1016/s0031-3955(05)70184-x. PMID 10629683
- [Background] Miller JL, Capino AC, Thomas A, Couloures K, Johnson PN. Sedation and Analgesia Using Medications Delivered via the Extravascular Route in Children Undergoing Laceration Repair. J Pediatr Pharmacol Ther. 2018 Mar-Apr;23(2):72-83. doi: 10.5863/1551-6776-23.2.72. PMID 29720907
- [Background] Ryan PM, Kienstra AJ, Cosgrove P, Vezzetti R, Wilkinson M. Safety and effectiveness of intranasal midazolam and fentanyl used in combination in the pediatric emergency department. Am J Emerg Med. 2019 Feb;37(2):237-240. doi: 10.1016/j.ajem.2018.05.036. Epub 2018 May 17. PMID 30146398
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kogan A, Katz J, Efrat R, Eidelman LA. Premedication with midazolam in young children: a comparison of four routes of administration. Paediatr Anaesth. 2002 Oct;12(8):685-9. doi: 10.1046/j.1460-9592.2002.00918.x. PMID 12472704
- [Background] Neville DN, Hayes KR, Ivan Y, McDowell ER, Pitetti RD. Double-blind Randomized Controlled Trial of Intranasal Dexmedetomidine Versus Intranasal Midazolam as Anxiolysis Prior to Pediatric Laceration Repair in the Emergency Department. Acad Emerg Med. 2016 Aug;23(8):910-7. doi: 10.1111/acem.12998. PMID 27129606